CLINICAL TRIAL: NCT06597890
Title: Move@NUS: Pilot Study of a Digital Intervention Cohort to Promote Healthy Sleep, Screen Viewing, and Physical Activity Habits for Improved Health and Wellbeing
Brief Title: Move@NUS: a Digital Intervention Cohort Promoting Healthy Movement Behaviours
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Dr Falk Mueller-Riemenschneider, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-800
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Inactivity; Sedentary Behavior; Sleep Insufficiency; Well-Being, Psychological
Keywords: smartphone; smartwatch; Apple Watch; ecological momentary assessment (EMA); ecological momentary intervention (EMI); mhealth; digital health
MeSH Terms: conditions — Sedentary Behavior; Sleep Deprivation; Psychological Well-Being | interventions — Organizational Objectives

STUDY DESIGN:
Intervention Model Description: 3x sequential 3-group randomised controlled trials (RCTs), embedded within the 6-month digital cohort study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- RCT 1 - group 1 (Experimental): Sleep Hygiene Ecological Momentary Intervention (EMI)
  Interventions: Behavioral: educational content (sleep hygiene); Behavioral: sleep hygiene strategies; Behavioral: reminders; Behavioral: review of behavioural goal; Behavioral: goal setting
- RCT 1 - group 2 (Experimental): Personalised Sleep Guideline EMI
  Interventions: Behavioral: reminders; Behavioral: review of behavioural goal; Behavioral: educational content (sleep guidelines); Behavioral: comparison of current behaviour to ideal behaviour; Behavioral: goal setting
- RCT 1 - group 3 (No Intervention): Control
- RCT 2 - group 1 (Experimental): Stair Climbing EMI
  Interventions: Behavioral: reminders; Behavioral: review of behavioural goal; Behavioral: comparison of current behaviour to ideal behaviour; Behavioral: goal setting
- RCT 2 - group 2 (Experimental): Vigorous Intermittent Lifestyle Physical Activity (VILPA) EMI
  Interventions: Behavioral: reminders; Behavioral: review of behavioural goal; Behavioral: goal setting; Behavioral: educational content (Vigorous Intermittent Lifestyle Physical Activity (VILPA))
- RCT 2 - group 3 (No Intervention): Control
- RCT 3 - group 1 (Experimental): Screentime Breaktime EMI
  Interventions: Behavioral: review of behavioural goal; Behavioral: comparison of current behaviour to ideal behaviour; Behavioral: screentime breaks
- RCT 3 - group 2 (Experimental): Screentime Goal EMI
  Interventions: Behavioral: reminders; Behavioral: review of behavioural goal; Behavioral: comparison of current behaviour to ideal behaviour; Behavioral: goal setting
- RCT 3 - group 3 (No Intervention): Control

INTERVENTIONS:
Behavioral: educational content (sleep hygiene) — app-based sleep hygiene-related educational content
  Arms: RCT 1 - group 1
Behavioral: sleep hygiene strategies — app-based self-selection of sleep hygiene strategies
  Arms: RCT 1 - group 1
Behavioral: reminders — daily reminders sent via push notifications
  Arms: RCT 1 - group 1; RCT 1 - group 2; RCT 2 - group 1; RCT 2 - group 2; RCT 3 - group 2
Behavioral: review of behavioural goal — app-based review of behavioural goal
  Arms: RCT 1 - group 1; RCT 1 - group 2; RCT 2 - group 1; RCT 2 - group 2; RCT 3 - group 1; RCT 3 - group 2
Behavioral: educational content (sleep guidelines) — app-based educational content on recommended sleep guidelines
  Arms: RCT 1 - group 2
Behavioral: comparison of current behaviour to ideal behaviour — use of smartwatch/smartphone data to assess current behaviour and compare it to ideal behaviour
  Arms: RCT 1 - group 2; RCT 2 - group 1; RCT 3 - group 1; RCT 3 - group 2
Behavioral: goal setting — prompt participant to set a goal in relation to targeted behaviour
  Arms: RCT 1 - group 1; RCT 1 - group 2; RCT 2 - group 1; RCT 2 - group 2; RCT 3 - group 2
Behavioral: educational content (Vigorous Intermittent Lifestyle Physical Activity (VILPA)) — app-based educational content on VILPA
  Arms: RCT 2 - group 2
Behavioral: screentime breaks — repeated daily reminders to break up screentime
  Arms: RCT 3 - group 1

SUMMARY:
The aim of the Move@NUS pilot study is to determine the feasibility of establishing a digital intervention cohort to monitor and improve the health and wellbeing of students by encouraging them to engage in healthy movement behaviours (i.e., physical activity, sleep, and limiting smartphone-based recreational screentime).

The digital intervention cohort consists of:

* 6-months of continuous monitoring of movement behaviours, wellbeing and related factors via an Apple Watch and repeated bursts of ecological momentary assessments (EMAs).
* 3x embedded randomised controlled trials (RCTs) evaluating the efficacy of small-scale smartphone-based interventions designed to nudge participants toward participating in healthier movement behaviours.

DETAILED DESCRIPTION:
Good overall mental and physical health and wellbeing can be promoted by engaging in healthy movement behaviours - getting adequate sleep, being physically active, and minimising recreational time spent watching a screen or being sedentary. The objectives of this study are to determine the feasibility of:

* establishing a digital cohort study and continuously monitoring health behaviours and wellbeing (and related factors) for 6 months, and
* rapidly evaluating the effects of ecological momentary interventions (EMIs; small-scale interventions that provide support in real-time, delivered via the smartwatch and app) for promoting healthy movement behaviours via a series of embedded RCTs.

The investigators will enrol up to 150 first-year university students into an innovative hybrid study that combines a digital cohort with embedded randomised controlled trials (RCTs). The digital cohort consists of 6 months of continuous observations of movement behaviours, wellbeing, and related factors via a smartwatch (Apple Watch) and repeated bursts of smartphone-based ecological momentary assessment (EMA) surveys. Throughout the 6-month monitoring period, participants are enrolled in 3 embedded RCTs evaluating the effects of EMIs that, in turn, target sleep, physical activity, and smartphone-based recreational screentime. For each embedded-RCT we assess engagement and acceptability outcomes (e.g., whether a push notification is opened, whether it is responded to), and preliminary efficacy (i.e., whether there is a between group difference in the target behaviour from pre- to post-intervention). Participants also complete traditional questionnaires at baseline, 3-, and 6-month follow-up.

ELIGIBILITY:
Participants are eligible to join the study if they:

* are enrolled in the first year of an undergraduate degree at the National University of Singapore,
* own or use an Apple smartphone with a data plan,
* are willing to download and use a smartphone app, and
* have an Apple smartwatch (Series 6/SE or newer) and are willing to wear it continuously for the 6-month study duration.

Participants will be excluded if they are:

* pregnant, or
* planning to be overseas for more than 6 weeks (per trip) during the upcoming semester.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
RCT 1. Sleep | week 1 (pre-intervention), week 3 (intervention midpoint), week 5 (post-intervention), and continuously throughout the 6-month study
  Sleep duration, as assessed via Apple Watch
RCT 2. Physical activity | week 6 (pre-intervention), week 8 (intervention midpoint), week 10 (post-intervention), and continuously throughout the 6-month study
  Step counts, as assessed via Apple Watch
RCT 2. Physical activity | week 6 (pre-intervention), week 8 (intervention midpoint), week 10 (post-intervention), and continuously throughout the 6-month study
  Flights of stairs climbed, as assessed via Apple Watch
RCT 2. Physical activity | week 6 (pre-intervention), week 8 (intervention midpoint), week 10 (post-intervention), and continuously throughout the 6-month study
  Moderate-to-vigorous physical activity, as assessed via Apple Watch
RCT 3. Screentime | week 6 (pre-intervention), week 8 (intervention midpoint), week 10 (post-intervention), and continuously throughout the 6-month study
  Screenshots of passively captured smartphone screentime data
Wellbeing | Continuously over 6-months
  Mental wellbeing, WHO-5 Well-Being Index (WHO-5; World Health Organisation). Min value 0, max value 100; higher scores indicate greater wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Falk Müller-Riemenschneider, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No